CLINICAL TRIAL: NCT01733849
Title: An Observational Study to Estimate the Disease Burden of Rotavirus Gastroenteritis in Infants/Children Less Than Five Years of Age in Primary Care Settings, in Bulgaria and Latvia
Brief Title: A Study to Estimate the Occurrence of Rotavirus Gastroenteritis in Children < 5 Years of Age, in Bulgaria and Latvia
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116621
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Infections, Rotavirus
Keywords: Bulgaria; Primary care settings; Children; Latvia; Acute gastroenteritis
MeSH Terms: conditions — Rotavirus Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group Bulgaria: Subjects in this group include infants/children from Bulgaria, less than five years of age with home visits by the GP/paediatrician for the treatment of AGE or brought to the GP/paediatrician for the treatment of AGE.
  Interventions: Other: Stool sample; Other: Data collection
- Group Latvia: Subjects in this group include infants/children from Latvia, less than five years of age with home visits by the GP/paediatrician for the treatment of AGE or brought to the GP/paediatrician for the treatment of AGE.
  Interventions: Other: Stool sample; Other: Data collection

INTERVENTIONS:
Other: Stool sample — Samples will be tested to determine the presence or absence of rotavirus.
Other: Data collection — Log books

SUMMARY:
This study aims to estimate the real situation of rotavirus gastroenteritis (RV GE) in the primary care settings of both Bulgaria and Latvia in children less than 5 years of age.

DETAILED DESCRIPTION:
A Primary care setting will include independent general practitioners (GP) (specialised in paediatrics) or independent paediatricians.

Stool samples will be collected from all enrolled subjects at Visit 1 (Day 0) and tested immediately after collection. The stool sample will be stored for 24 hours only, in case the test cannot be performed immediately after collection.

ELIGIBILITY:
Inclusion Criteria:

* Infants/children with home visits by the GPGP/paediatrician for the treatment of AGE or brought to the GP/paediatrician for AGE treatment during the study period.
* A male or female infant/child less than five years of age at the time of the GP/paediatrician visit. A child becomes ineligible on the day of her/his fifth birthday.
* Written informed consent obtained from the parents/legally acceptable representative (LARs) of the subject.
* Subjects who the investigator believes that his/her, parents/LARs can and will comply with the requirements of the protocol.

Exclusion Criteria:

• Child in care.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants/children less than five years of age with home visits by the GP/paediatrician for the treatment of AGE or brought to the GP/paediatrician for the treatment of AGE.
Sampling Method: Non-Probability Sample
Enrollment: 1266 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of RV GE cases among the acute gastroenteritis (AGE) cases reported at primary care settings in infants/children less than five years of age. | At the time of enrollment of each subject (Day 0).

SECONDARY OUTCOMES:
Symptoms related to AGE and their measures, stratified by rotavirus status for all the AGE cases reported by infants/children less than five years of age at the primary care settings. | Day 0 - Day 14+5 (At the time of phone call follow-up contact).
Number of RV GE cases reported at each month by infants/children less than five years of age reported at the primary care settings. | At the time of enrollment of each subject (Day 0).
Number of hospitalisations for RV GE and AGE, reported at the primary care settings. | At the time of phone call follow-up contact (14 to 19 days after enrollment).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (38):
- Bulgaria (11):
  - GSK Investigational Site, Burgas
  - GSK Investigational Site, Dobrich
  - GSK Investigational Site, Pazardzhik
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sliven
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Varna
  - GSK Investigational Site, Veliko Tarnovo
- Latvia (27):
  - GSK Investigational Site, Balvi
  - GSK Investigational Site, Bauska
  - GSK Investigational Site, Brocēni
  - GSK Investigational Site, Carnikava
  - GSK Investigational Site, Daugavpils
  - GSK Investigational Site, Druva
  - GSK Investigational Site, Erglu Pagasts
  - GSK Investigational Site, Grobiņa
  - GSK Investigational Site, Ikšķile
  - GSK Investigational Site, Jelgava
  - GSK Investigational Site, Jēkabpils
  - GSK Investigational Site, Kuldīga
  - GSK Investigational Site, Liepāja
  - GSK Investigational Site, Limbaži
  - GSK Investigational Site, Līvāni
  - GSK Investigational Site, Madona
  - GSK Investigational Site, Ogre
  - GSK Investigational Site, Ozolnieki
  - GSK Investigational Site, Piņķi
  - GSK Investigational Site, Rēzekne
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Ropaži
  - GSK Investigational Site, Sigulda
  - GSK Investigational Site, Tukums
  - GSK Investigational Site, Valmiera
  - GSK Investigational Site, Vangaži
  - GSK Investigational Site, Ventspils

REFERENCES:
- [Derived] Tafalla M, Gardovska D, Gopala K, Kozlovska L. Primary care-based surveillance to estimate the proportion of rotavirus gastroenteritis among Latvian children below 5 years of age with acute gastroenteritis. Hum Vaccin Immunother. 2019;15(6):1272-1278. doi: 10.1080/21645515.2018.1534515. Epub 2018 Oct 31. PMID 30335570
- [Derived] Tiholova M, Gopala K, Berberova M, Strokova-Stoilova M, Tafalla M. Rotavirus gastroenteritis in children less than five years of age in primary care settings in Bulgaria: an observational study. Germs. 2016 Sep 1;6(3):97-105. doi: 10.11599/germs.2016.1095. eCollection 2016 Sep. PMID 27622162